CLINICAL TRIAL: NCT07061743
Title: The Effect of Activity Management Training on Body Awareness, Cognitive Functions and Fatigue in Individuals With Chronic Low Back Pain
Brief Title: Activity Management Training in Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Nilay Şahan, Çankırı Karatekin University, Çankırı Karatekin University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8d4b4754e30644ac
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Low Back Pain
Keywords: Low back Pain, activity management training, cognitive function, fatique
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- low back pain group (Experimental)
  Interventions: Behavioral: activity management training

INTERVENTIONS:
Behavioral: activity management training — In activity management training, first week awareness training, second week ergonomics training, third week activity stepping training, fourth week joint-energy conservation training, and fifth week relaxation training will be given.

SUMMARY:
The individuals participating in the study will be asked to fill in the Body Awareness Scale, Canadian Activity Performance Measure, Pain Activity Patterns Scale, Cognitive Status Scale, and Fatigue Severity Scale. Afterwards, colour block design, puzzle making, and picture sorting subtests of the Loewenstein Occupational Therapy Cognitive Assessment will be applied to the individuals. After the initial assessments, activity management training will be provided to the patients. In the activity management training, first week awareness training, second week ergonomics training, third week activity stepping training, fourth week joint-energy conservation training, and fifth week relaxation training will be given. In the sixth and last week, the goals set will be reviewed. All pre-treatment tests will be re-administered at 6 weeks post-treatment. All applications will be carried out within Çankırı Karatekin University.

ELIGIBILITY:
Inclusion Criteria: literate individuals who have been complaining of low back pain for at least 3-6 months, who are willing to participate in the study -

Exclusion Criteria: Those with complaints of musculoskeletal pain due to cancer, fracture, or surgery in the last 6 months, those with serious psychiatric disorders such as panic disorder or major depression, and those who did not volunteer to participate in the study

-

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-07-03 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) | From enrollment to the end of treatment at 6 weeks
  The COPM is used to assess individuals' activity performance and satisfaction levels. In this assessment scale, the problems encountered by individuals in the field of activity performance are determined through a semi-structured interview. Individuals evaluate their activity performance problems with their own performance and satisfaction scores. In the first step, individuals are asked to identify the problems in the areas of self-care, productivity and leisure time that they do, want to do or have difficulty in doing in their routine. In the second step, individuals are asked to assign an importance value between 1 and 10 to each of these activities. In the third step, individuals are asked to select up to 5 activities that are most important for them and to give performance and satisfaction scores between 1 and 10 for each activity. The performance and satisfaction scores are totalled and divided by the number of activities to obtain performance and satisfaction scores.

SECONDARY OUTCOMES:
Body Awareness Questionnaire | From enrollment to the end of treatment at 6 weeks"
  The body awareness of the participants will be evaluated with the Body Awareness Questionnaire (BAQ) developed by Shields (31). The Turkish validity and reliability of the questionnaire was conducted by Karaca (2017). The questionnaire consists of four subscales (Note Changes in Response or Body Process, Predict Body Response, Onset of Illness, and Sleep-Wake Cycle) and 18 questions in total. The questionnaire is scored on a 7-point Likert scale ranging from 'Not true for me' (1) to 'Completely true for me' (7).
Pain Activity Patterns Scale (PAPS) | From enrollment to the end of treatment at 6 weeks
  The PAPS is a scale that determines the changing activity patterns in individuals with chronic pain in 3 subgroups as avoidance, excessive avoidance and regularisation. It was developed by Cane et al. in Canada. The AAPS consists of 3 subgroups, including avoidance, excessive avoidance, and regularisation, and a total of 30 questions, 10 for each subgroup. In the scale, individuals with chronic pain are asked to answer questions about how they perform activities of daily living. In answering the questions in the scale, a 5-point Likert scoring system is used, 0-never, 2-sometimes, 4-always. In the calculation of the scale score, separate score calculations are made for the subgroups of avoidance, overdoing, and regularisation. The total scores calculated for the subgroups vary between 0-40 points separately. Within these 3 subgroups, the subgroup with the highest score by the patient is determined and it is determined which subgroup the participant adopts in activities of daily living
Loewenstein Occupational Therapy Cognitive Assessment (LOTCA) | From enrollment to the end of treatment at 6 weeks
  The Loewenstein Occupational Therapy Cognitive Assessment (LOTCA) will be used in the study to evaluate the basic cognitive skills of individuals. The test consists of 22 items, including 2 items of orientation, 6 items of visual-spatial perception, 7 items of visual-motor organisation, 6 items of thinking skills, and 1 item of attention. The content of the test (36): Orientation: 1. Time orientation 2. Place orientation Visual perception: 1. object recognition 2. shape recognition 3. overlapping figures 4. object invariance 5. spatial perception 6. praxis Visual-motor organisation: 1. Geometric shape copying 2. Two-dimensional model 3. Pegboard construction 4. Coloured block design 5. Plain block design 35 6. Jigsaw puzzle 7. Clock drawing Thinking Skills: 1. Categorisation 2. Risca Object Classification I - structured (Risca Object Classification- ROC I) 3. Riska Object Classification II - unstructured (ROC II) 4. Picture Sorting A 5. Picture Sorting B 6. Geometric Sorting Attention
Stroop test | From enrollment to the end of treatment at 6 weeks
  The Stroop Test is a neuropsychological test that reflects frontal region activity. It measures the brain's ability to direct attention, conceptual flexibility and mental processing speed. In the first stage of the Stroop attention test, people are presented with the names of colours and asked to read these colours quickly. For example, no matter what colour the font is, it will be read as 'red'. In the second step, they are asked to quickly say what colour the dot clusters printed through ink are. For example, if the word 'red' is written in yellow font, they should say "yellow" instead of 'red'. In the final stage of the test, the third stage, the participants are asked to say the words written in a different colour than the name of the colour as fast as possible in a loud voice. For example, the word 'blue' is written in red or black. As a result of these experiments, the Stroop effect occurs. When it was investigated with imaging techniques where the Stroop effect affects the hum
Cognitive Status Scale | From enrollment to the end of treatment at 6 weeks
  It was developed by Broadbent et al. to assess cognitive failures that occur in daily life. Failures in perception, memory, and motor functions are assessed with 25 questions. Each question is scored between 0 (never) and 4 (very often) in the scale consisting of questions such as 'Do you ever find yourself accidentally hiding what you should throw away and throwing away what you should keep?', 'Do you ever forget people's names?', 'Do you drop things?'. The total score ranges from 0-100, with a higher score indicating an increased level of cognitive failure. The validity and reliability study of the Turkish version of the scale was conducted by Ekici et al.
Fatigue Severity Scale | From enrollment to the end of treatment at 6 weeks
  The scale was developed by Krup et al. (1989), and its Turkish validity and reliability were examined by Armutlu et al. (2007). The scale has 9 questions and one dimension. The individual indicates the level of agreement with the items in the scale by choosing a number from 1 (strongly disagree) to 7 (strongly agree). A total score of 9-63 can be obtained from the scale. A total score of 36 or more indicates severe fatigue

CONTACTS AND LOCATIONS:
Locations (1):
- Çankırı Karatekin University, Çankırı, Uluyazı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No